CLINICAL TRIAL: NCT05259592
Title: Patient-centered Modular Cognitive Behavioral Therapy for Complex PTSD: A Randomised Controlled Pilot Study
Brief Title: Patient-centered Modular CBT for CPTSD: A Randomised Controlled Pilot Study
Acronym: PACE pilot RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Danish Veterans Centre (Other Government)
Collaborators: University of Copenhagen (Other); Edinburgh Napier University (Other)
Responsible Party: Principal Investigator, Sofie Folke, Principal Investigator, Danish Veterans Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-871
Record Dates: First submitted 2022-01-19; First posted 2022-02-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Complex Post-Traumatic Stress Disorder
Keywords: CBT; Modular therapy; pilot randomized controlled study
MeSH Terms: conditions — Color Vision Defects | interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study is a randomised controlled pilot study that follows the guidelines of the Consolidated Standards of Reporting Trials (CONSORT; Boutron et al., 2017) and the SPIRIT guidelines (Chan et al., 2013).
  60 Danish veterans with complex PTSD (CPTSD) will be randomised to either modular patient-centred CBT (MPC) or a control treatment, where the order of the treatment modules is determined in advance. A randomisation list was prepared using R software (www.r-project.org). Participants are randomised into the intervention group or the control group with 30 participants in each group, stratified by recruitment/treatment site. A block size of six will be used to ensure an even balance. The randomisation was pre-pared by a data manager affiliated with the project, and only he is able to see the randomisation list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modular Patient Centred CBT (MPC) for CPTSD (Experimental): MPC (Folke, Friis, Thomsen & Roitmann, 2020) is a treatment programme consisting of up to 32 therapy sessions broken down by five treatment modules (each consisting of six sessions). Prior to the treatment modules, the client completes an intro module (two sessions) focusing on psyhoeducation on CPTSD, individual case formulation and introduction to the further treatment programme. After the intro module (and after each treatment module), the client and therapist jointly decide which treatment module to proceed with based on 'co-decision'. The treatment modules directly address the symptoms of CPTSD: 1) Affect dysregulation, 2) Disturbed relationships, 3) Negative self-concept, 4) PTSD symptoms, and 5) Insomnia and trauma-related nightmares. Each treatment module is structured in such a way that it can be offered alone and independently of the other modules.
  Interventions: Behavioral: Psychotherapy
- Modular CBT for CPTSD without co-decision (Active Comparator): Because the study investigates a potentially beneficial effect of including the client directly in treatment decisions (by having the client determine the order of treatment modules together with the therapist), the patient-centred version of the treatment is compared with a control treatment, where the five treatment modules are delivered in a predefined order. The control treatment thus consists of the same treatment components as described above. It is only the aspect of co-decision that has been taken out. Instead, the therapist will just inform the client about the order of treatment modules in the programme. The order of treatment modules in the control treatment will be: 1) Affect dysregulation (6 sessions), 2) Disturbed relationships (6 sessions), 3) Negative self-concept (6 sessions), 4) PTSD symptoms (6 sessions) and 5) Insomnia and trauma-related nightmares (6 sessions).
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Modular Patient Centred CBT (MPC) for CPTSD (Folke, Friis, Thomsen & Roitmann, 2020) is a psychotherapy treatment manual consisting of up to 32 individual therapy sessions broken down by five treatment modules (each consisting of six sessions) that directly address the symptoms of CPTSD: 1) Affect dysregulation, 2) Disturbed relationships, 3) Negative self-concept, 4) PTSD symptoms, and 5) Insomnia and trauma-related nightmares.

SUMMARY:
Modular Patient Centred CBT (MPC) for Complex PTSD (CPTSD) is a manualized psychotherapy programme that consists of five treatment modules addressing 1) Affect dysregulation, 2) Disturbed relationships, 3) Negative self-concept, 4) PTSD symptoms and 5) Insomnia and trauma-related nightmares.

This aim of this first pilot randomised controlled trial (RCT) is to increase chances of a future successful efficacy RCT (Phase III trial) comparing the efficacy (on symptoms of CPTSD and co-morbid disorders) of a flexible, patient-centred version of the MPC treatment programme (where the client actively participates in treatment decisions) with a control treatment, where the five treatment modules are delivered in a predefined order.

The primary objective of the pilot study is to:

1. Assess the implementation of the trial process in terms of inclusion, implementation and data collection
2. Assess necessary resources, including the use of tablets for data collection, time spent on the project by participating therapists, assessing psychologists and secretaries

The secondary objective is to:

1. Assess changes in symptoms of CPTSD between the intervention and control group as well as within each group
2. Examine changes in levels of comorbidity associated with CPTSD, such as anxiety, depression, insomnia, somatic complaints, drugs and alcohol intake between the intervention and control group as well as within each group
3. Examine changes in well-being, functioning and attachment style between the intervention and control group as well as within each group
4. Examine developments in client motivation and working alliance between the intervention and control group as well as within each group.

60 veterans with CPTSD are randomised to receive either the flexible, patient-centred version of the MPC treatment programme or the control treatment.

The investigators will consider the study as complete if the following success criteria are met:

1. > 70% of potential participants accept and be included in the study
2. Completion rate of 70%, that is, the investigators expect to have complete end-of-treatment data of at least 70% of all participants included
3. Complete three-month follow-up of at least 50% of all participants included.

The project neither collects new biological material nor biological material from existing biobanks. The project is based on questionnaire data.

DETAILED DESCRIPTION:
ICD-11 complex PTSD (CPTSD) is a new diagnosis and up to this date, no effective treatment has been identified to help clients with this severe mental disorder. Therefore, it is very important that effective treatment methods for clients with CPTSD be identified.

In 2019 the Danish Veteran Centre launched the development of a treatment programme for veterans with CPTSD; Modular Patient Centred CBT (MPC) for CPTSD. MPC is a manualised treatment programme that consists of 32 individual psychotherapy sessions, divided into an initial treatment module (two therapy sessions) and five treatment modules (each consisting of six therapy sessions) that can be combined in different ways to adapt to each client's most prominent symptoms, preferences and readiness (to work with exposure, for instance). The five treatment modules address 1) Affect dysregulation (6 sessions), 2) Disturbed relationships (6 sessions), 3) Negative self-concept (6 sessions), 4) PTSD symptoms (6 sessions) and 5) Insomnia and trauma-related nightmares (6 sessions).

This first trial of the MPC treatment programme is conducted as a pilot randomised controlled trial. The primary objective of this study is to increase chances of a future successful efficacy RCT (Phase III trial) comparing the efficacy (on symptoms of CPTSD and co-morbid disorders) of a flexible, patient-centred version of the MPC treatment programme (where the client actively participates in treatment decisions) with a control treatment, where the five treatment modules are delivered in a predefined order; 1) Affect dysregulation, 2) Disturbed relationships, 3) Negative self-concept, 4) PTSD symptoms, and 5) Insomnia and trauma-related nightmares.

The primary objective of the pilot study is to:

1. Assess the implementation of the trial process in terms of inclusion, implementation and data collection
2. Assess necessary resources, including the use of tablets for data collection, time spent on the project by participating therapists, assessing psychologists and secretaries

The secondary objective is to:

1. Assess changes in symptoms of CPTSD, assessed with the International Trauma Questionnaire (ITQ; Cloitre et al., 2018) between the intervention and control group as well as within each group
2. Examine changes in levels of comorbidity associated with CPTSD, such as anxiety, depression, insomnia, somatic complaints, drugs and alcohol intake between the intervention and control group as well as within each group
3. Examine changes in well-being, functioning and attachment style between the intervention and control group as well as within each group
4. Examine developments in client motivation and working alliance between the intervention and control group as well as within each group.

60 veterans with CPTSD are randomised to receive either the flexible, patient-centred version of the MPC treatment programme or the control treatment. As an integral part of the treatment, a short assessment is conducted after each treatment module by having the client complete the primary outcome measure, the ITQ which is used as a measure for assessing ICD-11 PTSD and CPTSD. In practice, the client fills in the ITQ on a tablet in the beginning of the last session of each treatment module, after which the client and therapist receive an automatic response on the tablet, establishing whether the client (based on the ITQ) continues to meet the diagnostic criteria for PTSD or CPTSD. If the client has achieved sufficient symptom recovery and no longer meets the diagnostic criteria for CPTSD, the client is considered a treatment completer. However, the client and the therapist might decide to continue treatment until the client no longer meets the diagnostic criteria for PTSD. In this way, treatment can continue to up till 32 therapy sessions but client and therapist can end the treatment earlier if the client has a valid assessment and falls out of CPTSD criteria.

Since the study is a pilot study, aiming to inform a future RCT, the investigators will consider the study as complete if the following success criteria are met:

1. > 70% of potential participants accept and be included in the study
2. Completion rate of 70%, that is, the investigators expect to have complete data (end-of-treatment outcome assessment completed at the final therapy session) of at least 70% of all participants included
3. Complete three-month follow-up of at least 50% of all participants included.

The treatment is carried out at five local veteran centres in Denmark by clinical psychologists employed by the Military Psychology Department (MPD), Danish Veterans Centre. The participating psychologists receive training and regular method-specific supervision in the MPC treatment programme.

The project neither collects new biological material nor biological material from existing biobanks. The project is based on questionnaire data

Note regarding study objectives, results reporting, and start date (added March 2025):

The original registration emphasized feasibility-related objectives as primary, including aspects of recruitment, implementation, and data collection. Clinical outcomes listed as secondary objectives have also been explored in more depth in the final analyses and will be reported in a forthcoming manuscript.

As this study does not qualify as an Applicable Clinical Trial (ACT) under FDAAA 801, results submission is not required by law. However, results will be submitted voluntarily after acceptance of the primary publication to ensure transparency and consistency with journal embargo policies.

The Study Start Date was also updated to January 5, 2021, to reflect the actual date of first participant enrollment with completed baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for CPTSD, assessed with the ITQ
* Danish veteran (cf. the Veteran Policy of Denmark )
* Seeks help at the Military Psychology Department, Danish Veterans Centre, for deployment-related psychological issues

Exclusion Criteria:

* Severely suicidal
* Current alcohol or drug abuse that prevents treatment
* Blast injuries or current severe attention disorder
* Has received psychotherapeutic treatment in the past three months
* Is participating in another research project that interferes with this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
The International Trauma Questionnaire (ITQ; Cloitre et al., 2018) | Through study completion, up to 1 year
  20-item self-report scale that assesses the diagnostic criteria for PTSD and CPTSD according to ICD-11

SECONDARY OUTCOMES:
The Insomnia Severity Index (ISI) | Through study completion, up to 1 year
  7-item self-report scale that assesses insomnia
The Depression Anxiety Stress Scales (DASS-42) | Through study completion, up to 1 year
  42-item self-reporting instrument designed to measure three related negative emotional stages of depression, anxiety and tension/stress
Item 1-12 from the Common Mental Disorders Questionnaire (CMDQ) | Through study completion, up to 1 year
  12 item self-report scale that assesses somatic symptoms
3 items from the Alcohol Use Disorders Identification Test (AUDIT). | Through study completion, up to 1 year
  Three questions about alcohol consumption; 1) how often the client consumes alcohol; 2) how many items the client consumes on a typical day, and 3) whether the client has been treated for alcohol abuse.
7 items on cannabis and other forms of drugs | Through study completion, up to 1 year
  Questions on cannabis and other forms of drugs. The questions have previously been used in surveys by the Danish Veteran Centre and the National Institute of Public Health, the University of Southern Denmark.
World Health Organization Well-being Index (WHO-5) | Through study completion, up to 1 year
  5 item self-report scale that assesses subjective psychological well-being
The Sheehan Disability Scale (SDS) | Through study completion, up to 1 year
  3 item self-report scale that assesses occupational, social and family functioning
The Experiences in Close Relationships - Short form (ECR-S) | Through study completion, up to 1 year
  12 item self-report scale that assesses adult attachment style

CONTACTS AND LOCATIONS:
Overall Officials: Sofie Folke, PhD, Principal Investigator — Military Psychology Department, Danish Veteran Centre
Locations (5):
- Denmark (5):
  - Danish Veterans Centre, Aalborg Kaserner, Aalborg
  - Danish Veterans Centre, Garderkasernen, Birkerød
  - Danish Veterans Centre, Svanemoellen Kaserne, Copenhagen Ø
  - Danish Veterans Centre, Ryes Kaserne, Fredericia
  - Danish Veterans Centre; Ringsted Kaserne, Ringsted

IPD SHARING:
Plan to Share IPD: No
Due to privacy and data protection regulations of the Danish Defence, data from the current study cannot be shared.

REFERENCES:
- [Background] Folke, S, Friis, K, Thomsen, U, & Roitmann, N. Modulopbygget Patient-centreret CBT til Kompleks-PTSD - behandlingsmanual version 1.0. Unpublished manual. 2020
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT05259592/Prot_SAP_000.pdf